CLINICAL TRIAL: NCT06611514
Title: Effect of Intravaginal Prasterone on Genitourinary Syndrome in Women in Menopause With Previous Breast Cancer or Currently Under Treatment With Endocrine Therapy for Breast Cancer With Aromatase Inhibitor +/- LHRHa
Brief Title: Effect of Intravaginal Prasterone on Symptoms of Genitourinary Syndrome of Menopause (GSM) in Women in Menopause With Previous Breast Cancer
Acronym: PROPOSE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UID 2966
Record Dates: First submitted 2024-09-12; First posted 2024-09-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-09

CONDITIONS: Women With Breast Cancer
Keywords: genitourinary syndrome; prasterone; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intravaginal Prasterone (Experimental)
  Interventions: Drug: Prasterone (DHEA)

INTERVENTIONS:
Drug: Prasterone (DHEA) — Prasterone 6.5 mg vaginal tablets

SUMMARY:
The goal of this interventional study is to evaluate the effect of Intravaginal Prasterone for the treatment of moderate to severe symptoms of genitourinary syndrome (GSM) due to natural, surgical or treatment-induced menopause and the effect on the quality of life, including sexual function and mood well-being, in women with Breast Cancer. A sample size of 95 patients will be needed to show that the proportion of women showing symptom improvement is greater than 50%. Subjects will be followed up at four weeks and twelve weeks of treatment. One and three-month outcomes will be provided after the end of treatment. Comparison between menopausal women with previous breast cancer that have finished hormonal therapy or with ER negative breast cancer and women currently under endocrine therapy with AIs will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer, completely excised
* Natural or iatrogenic menopausal status
* No evidence of distant metastasis
* Self-identified moderate to severe symptoms of genitourinary syndrome
* Normal kidney and liver function
* Written Informed Consent signed and dated by patient
* Negative Papanicolau (Pap) Smear Cytology Test within 1 year prior to enrollment

Exclusion Criteria:

* Vaginal or uterine bleeding of unknown origin
* Current diagnosis of any non-breast malignancy
* Metastatic disease
* Currently on chemiotherapy
* Currently on treatment with tamoxifen
* Mentally incompetent or evidence of active substance or alcohol abuse
* Endometrial hyperplasia
* Pregnancy or lactation
* Currently use of other vaginal therapy for the same purpose (if present, they have to be stopped 15 days before baseline visit)
* Clinically significant metabolic or endocrine disease not controlled by medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Establish subjective improvement in genitourinary symptomatology at intervals marked by the study | From enrollment to after 3 months after the end of treatment
  To establish the improvement in vulvovaginal and urinary symptoms, by subjective evaluation at baseline, at 12 weeks and after 1 and 3 months after the end of the treatment. Establish tissue trophism improvement through gynecological evaluation, the use of validated scales (Vaginal Health Index), and determination of the maturation index on vaginal spatula, measure serum estradiol during and after treatment
evaluation of vulvovaginal and urinary symptoms | 6 months
  evaluation of vaginal dryness, dyspareunia, pruritis, burning and dysuria with a 0 to 4 score (0: absence, 1: mild, 2: moderate, 3: severe, 4: very severe)
improvement in vaginal signs | 6 months
  To establish the improvement in vaginal signs using the Vaginal Health Index Scale (VHI)
evaluation fo maturation index | 6 months
  To assess the maturation index (as percentage of superficial, intermediate and parabasal cells) in the vaginal mucosa
grade of satisfaction | 6 months
  To report the grade of satisfaction as measured by the Global Response Assessment at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: SILVIA MARTELLA, Principal Investigator — European Institue of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy